CLINICAL TRIAL: NCT03194789
Title: The Effect of Footwear Generated Biomechanical Manipulation on Symptoms of Stress Urinary Incontinence
Acronym: SUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-7163
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Floor Disorders; Stress Urinary Incontinence
Keywords: FGBMM; LPSE; UDI - 6; UIQ - 7
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Single blinded (evaluator), single-center, randomized controlled trial Interventional and Control group.
Who Masked: Outcomes Assessor
Masking Description: Randomized single blinded (evaluator) controlled trial. The outcomes assessor will be masked in the study. Assessor will be independent of randomization, trial coordination and care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional Pelvic Floor Therapy (Active Comparator): up to six sessions, with one session every alternate week.
  Interventions: Other: Traditional Pelvic Floor Therapy
- FGBMM plus Traditional pelvic floor therapy (Experimental): Treatment with FGBMM using shoes with pertupods daily at home along with traditional pelvic floor therapy sessions.
  Interventions: Device: Footwear Generated Bio-Mechanical Manipulation (using shoes with pertupods) along with Traditional Pelvic Floor Therapy

INTERVENTIONS:
Device: Footwear Generated Bio-Mechanical Manipulation (using shoes with pertupods) along with Traditional Pelvic Floor Therapy — Participants will have FGBMM using shoes with pertupods along with traditional pelvic floor therapy over the course of six months. This will include five sessions of gait assessment and re-calibration with daily at home exercise with the device (shoes) over the course of six months. Along with that, participant will receive traditional pelvic floor therapy of six sessions, up-to one sessions every alternate week. This will involve exercise and modalities as decided by medical providers and therapists. Participants will also have a home exercise program prescribed along with each session and for the remainder of six months.
  Arms: FGBMM plus Traditional pelvic floor therapy
Other: Traditional Pelvic Floor Therapy — Participant will receive traditional pelvic floor therapy of six sessions, up-to one sessions every alternate week. This will involve exercise and modalities as decided by medical providers and therapists. Participants will also have a home exercise program prescribed along with each session and for the remainder of six months.
  Arms: Traditional Pelvic Floor Therapy

SUMMARY:
FGBMM (footwear generated biomechanical manipulation) effects neuromuscular patterns of pelvic muscles. While there have been no published studies to our knowledge investigating the effect of FGBMM on urinary incontinence, FGBMM causes perturbations in balance and gait that create dynamics similar to dynamic lumbosacral stabilization exercises. The investigators propose that FGBMM induces the same bio-mechanical improvements as LPSE (lumbopelvic stabilization exercises) which have shown benefit for incontinence. Instead of instructing patients to co-contract the lower trunk and pelvic floor muscles as commonly done for LPSE, the shoes used in FGBMM can be calibrated in a way that causes this co-contraction to occur without the patient realizing. Beneficial pelvis and spine positioning can also be accomplished by strategic placement of the pods without having to instruct the patient on complicated maneuvers. Capitalizing on the excellent adherence and clinical benefits of FGBMM on related conditions, the investigators propose to evaluate the effects of FGBMM in addition to pelvic floor therapy for improving the symptoms of stress urinary incontinence in an urban inner city population.

DETAILED DESCRIPTION:
FGBMM (footwear generated biomechanical manipulation) effects neuromuscular patterns of pelvic muscles. While there have been no published studies to our knowledge investigating the effect of FGBMM on urinary incontinence, FGBMM has been shown to cause perturbations in balance and gait that create dynamics similar to dynamic lumbosacral stabilization exercises. In support of this theory, although not published, one of the founders of the technique, Avi Elbaz, has noted anecdotal evidence that patients who had SUI (stress urinary incontinence) and underwent FGBMM for knee or low back pain reported improvement of incontinence. The investigators propose that FGBMM induces the same bio-mechanical improvements as LPSE (lumbopelvic stabilization exercises) which have shown benefit for incontinence. The pods on the footwear can be positioned to challenge the patients balance in a manner similar to the way trampolines are utilized in LPSE. Instead of instructing patients to co-contract the lower trunk and pelvic floor muscles as commonly done for LPSE, the shoes used in FGBMM can be calibrated in a way that causes this co-contraction to occur without the patient realizing. Beneficial pelvis and spine positioning can also be accomplished by strategic placement of the pods without having to instruct the patient on complicated maneuvers. An additional advantage of FGBMM is that this exercise is done with increased intra-abdominal pressure mimicking the condition and the setting when incontinence occurs rather than static exercise that is used in PFT. While performing regular activities, people are naturally squatting and doing other activities that increase intra-abdominal pressure. Furthermore, FGBMM is more practical for people with busy schedules because it can be accomplished with a much smaller time commitment from the patient than traditional PFT since it is done during normal activity. Capitalizing on the excellent adherence and clinical benefits of FGBMM on related conditions, the investigators propose to evaluate the effects of FGBMM in addition to pelvic floor therapy for improving the symptoms of stress urinary incontinence in an urban inner city population.

A potential use of FGBMM using shoes as a addition to traditional pelvic floor therapy may yield a more effective therapy with better adherence. Problems with traditional therapy include poor patient adherence (patients often do not complete the sessions and have poor adherence (about 50%), lack of the continuation in an ongoing program, leading to relapse and need for re treatment or even little clinical benefit. Additionally, access to pelvic floor therapy is limited for many patients since there are not enough available outpatient therapy services to meet the needs of all patients. Finding an additional exercise program that will increase adherence and improve patient outcomes with better clinical benefits is a high priority from both patient care and cost management perspectives.

FGBMM using shoes potentially overcomes many of these issues with improving/modifying abnormal biomechanics of pelvic floor muscles (therefore decreasing incontinence), and a home based exercise program utilizing footwear that causes exercise with normal activity by promoting perturbation. This bio-mechanical approach may significantly improve the symptoms of urinary incontinence in patients with Stress SUI or Mixed urinary incontinence. Capitalizing on the reported excellent adherence and clinical benefit of FGBMM in patients with related conditions, the investigators propose to evaluate the bio-mechanical exercise (wearing an appropriately calibrated shoe at home for a prescribed amount of time each day) as a conservative treatment that may supplement traditional pelvic floor therapy, medications and even surgical intervention for the same in an inner urban city population.

ELIGIBILITY:
Inclusion Criteria:

* Stress or Mixed Urinary Incontinence, based on UDI-6.
* Females between the ages of 18-75 years.
* Weight less than 350 lbs.
* Ambulatory and active patients that can participate in a rehabilitation program that includes daily walking
* Able to walk at least 50 meters and scored positive on the STEADI test
* Able to understand, read and sign the informed consent form
* English or Spanish speaking

Exclusion Criteria:

* Prior surgery for incontinence
* Pelvic Floor Therapy within past 6 months.
* Currently pregnant
* Predominantly Urge Incontinence.
* Patients with more than 3 falls in the last 52 weeks, OR any balance related fall with an injury in the last 52 weeks.
* Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedure.
* Patients with a history of pathological osteoporotic fracture
* Any major cardiovascular comorbidities prohibiting enrollment in an active exercise program
* Active heart disease (ischemia or heart failure admissions within 24 weeks) and Active COPD (exacerbation within 24 weeks)
* Active malignancies on ongoing treatment
* Patient with neurological gait pattern.
* Patient requiring assistive device during gait analysis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators traditionally see stress urinary incontinence patients, most commonly females, in our clinics everyday. The investigators only have about one patient visit per month in our clinics as 'males with same disorder.' To get a significant number of male patients in our study with the same condition will need at least 7-10 years approximately.
Enrollment: 55 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Severity of Stress Urinary Incontinence | Six months
  Improvement in symptoms of Stress Urinary Incontinence (SUI) measured by Urinary Distress Inventory) UDI - 6 questionnaire

SECONDARY OUTCOMES:
Quality of Life as determined by the Urinary Impact Questionnaire (UIQ-7) | Six months
  Change in Quality of Life from baseline will be determined with the use of the UIQ-7 questionnaire. Specifically, the UIQ-7 questionnaire is used to measure the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions. The UIQ-7 is a subscale of the PFIQ-7 and consists of 7 questions related to urinary symptoms and its effect on function, social health, and mental health. Responses for each question range from 0 (=not at all) to 3 (=quite a bit). Scores are summarized. A lower score indicates less impact on quality of life based on urinary symptoms.
Pelvic Floor Muscle Activity | Six months
  Assessment of Pelvic Floor Muscle Activity by surface EMG (electromyography)
Gait assessment | Six months
  Objective assessment of patient's gait measured by gait analysis equipment.
Adherence to treatment | Six months
  Compliance to FGBMM and PFT using questionnaire.
6 minute walk test | Six months
  objective assessment using maximum distance comfortably walked in 6 minutes on a 100 foot closed course
Medication costs | six months
  changes in medication costs assessed by patient interview
Healthcare utilization | six months
  Changes in healthcare facility utilization assessed by patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Lasak, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center - Medical Park Campuses, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng K, Cheung RYK, Lee LL, Chung TKH, Chan SSC. An observational follow-up study on pelvic floor disorders to 3-5 years after delivery. Int Urogynecol J. 2017 Sep;28(9):1393-1399. doi: 10.1007/s00192-017-3281-z. Epub 2017 Feb 14. PMID 28197646
- [Background] de Souza Abreu N, de Castro Villas Boas B, Netto JMB, Figueiredo AA. Dynamic lumbopelvic stabilization for treatment of stress urinary incontinence in women: Controlled and randomized clinical trial. Neurourol Urodyn. 2017 Nov;36(8):2160-2168. doi: 10.1002/nau.23261. Epub 2017 Mar 27. PMID 28346721
- [Background] Barzilay Y, Segal G, Lotan R, Regev G, Beer Y, Lonner BS, Mor A, Elbaz A. Patients with chronic non-specific low back pain who reported reduction in pain and improvement in function also demonstrated an improvement in gait pattern. Eur Spine J. 2016 Sep;25(9):2761-6. doi: 10.1007/s00586-015-4004-0. Epub 2015 May 16. PMID 25981205
- [Background] Ghaderi F, Mohammadi K, Amir Sasan R, Niko Kheslat S, Oskouei AE. Effects of Stabilization Exercises Focusing on Pelvic Floor Muscles on Low Back Pain and Urinary Incontinence in Women. Urology. 2016 Jul;93:50-4. doi: 10.1016/j.urology.2016.03.034. Epub 2016 Apr 5. PMID 27059833
- [Background] Silva VR, Riccetto CL, Martinho NM, Marques J, Carvalho LC, Botelho S. Training through gametherapy promotes coactivation of the pelvic floor and abdominal muscles in young women, nulliparous and continents. Int Braz J Urol. 2016 Jul-Aug;42(4):779-86. doi: 10.1590/S1677-5538.IBJU.2014.0580. PMID 27564290
- [Background] Solomonow-Avnon D, Levin D, Elboim-Gabyzon M, Rozen N, Peled E, Wolf A. Neuromuscular response of hip-spanning and low back muscles to medio-lateral foot center of pressure manipulation during gait. J Electromyogr Kinesiol. 2016 Jun;28:53-60. doi: 10.1016/j.jelekin.2016.02.010. Epub 2016 Mar 9. PMID 27016625
- [Background] Tahtinen RM, Cartwright R, Tsui JF, Aaltonen RL, Aoki Y, Cardenas JL, El Dib R, Joronen KM, Al Juaid S, Kalantan S, Kochana M, Kopec M, Lopes LC, Mirza E, Oksjoki SM, Pesonen JS, Valpas A, Wang L, Zhang Y, Heels-Ansdell D, Guyatt GH, Tikkinen KAO. Long-term Impact of Mode of Delivery on Stress Urinary Incontinence and Urgency Urinary Incontinence: A Systematic Review and Meta-analysis. Eur Urol. 2016 Jul;70(1):148-158. doi: 10.1016/j.eururo.2016.01.037. Epub 2016 Feb 10. PMID 26874810
- [Background] Utomo E, Korfage IJ, Wildhagen MF, Steensma AB, Bangma CH, Blok BF. Validation of the Urogenital Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7) in a Dutch population. Neurourol Urodyn. 2015 Jan;34(1):24-31. doi: 10.1002/nau.22496. Epub 2013 Oct 26. PMID 24167010
- [Background] Bush HM, Pagorek S, Kuperstein J, Guo J, Ballert KN, Crofford LJ. The Association of Chronic Back Pain and Stress Urinary Incontinence: A Cross-Sectional Study. J Womens Health Phys Therap. 2013 Jan;37(1):11-18. doi: 10.1097/JWH.0b013e31828c1ab3. PMID 23794961
- [Background] Timmermans L, Falez F, Melot C, Wespes E. Validation of use of the International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF) for impairment rating: a transversal retrospective study of 120 patients. Neurourol Urodyn. 2013 Sep;32(7):974-9. doi: 10.1002/nau.22363. Epub 2012 Dec 31. PMID 23281067
- [Background] Hides J, Stanton W, Mendis MD, Sexton M. The relationship of transversus abdominis and lumbar multifidus clinical muscle tests in patients with chronic low back pain. Man Ther. 2011 Dec;16(6):573-7. doi: 10.1016/j.math.2011.05.007. Epub 2011 Jun 8. PMID 21641268
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Eliasson K, Elfving B, Nordgren B, Mattsson E. Urinary incontinence in women with low back pain. Man Ther. 2008 Jun;13(3):206-12. doi: 10.1016/j.math.2006.12.006. Epub 2007 Mar 23. PMID 17363318
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Hajebrahimi S, Corcos J, Lemieux MC. International consultation on incontinence questionnaire short form: comparison of physician versus patient completion and immediate and delayed self-administration. Urology. 2004 Jun;63(6):1076-8. doi: 10.1016/j.urology.2004.01.005. PMID 15183953
- [Background] Sapsford R. Rehabilitation of pelvic floor muscles utilizing trunk stabilization. Man Ther. 2004 Feb;9(1):3-12. doi: 10.1016/s1356-689x(03)00131-0. PMID 14723856
- [Background] Fultz NH, Burgio K, Diokno AC, Kinchen KS, Obenchain R, Bump RC. Burden of stress urinary incontinence for community-dwelling women. Am J Obstet Gynecol. 2003 Nov;189(5):1275-82. doi: 10.1067/s0002-9378(03)00598-2. PMID 14634553
- [Background] van der Vaart CH, de Leeuw JR, Roovers JP, Heintz AP. Measuring health-related quality of life in women with urogenital dysfunction: the urogenital distress inventory and incontinence impact questionnaire revisited. Neurourol Urodyn. 2003;22(2):97-104. doi: 10.1002/nau.10038. PMID 12579625
- [Background] Persson J, Wolner-Hanssen P, Rydhstroem H. Obstetric risk factors for stress urinary incontinence: a population-based study. Obstet Gynecol. 2000 Sep;96(3):440-5. doi: 10.1016/s0029-7844(00)00950-9. PMID 10960639
- [Background] Brown JS, Grady D, Ouslander JG, Herzog AR, Varner RE, Posner SF. Prevalence of urinary incontinence and associated risk factors in postmenopausal women. Heart & Estrogen/Progestin Replacement Study (HERS) Research Group. Obstet Gynecol. 1999 Jul;94(1):66-70. doi: 10.1016/s0029-7844(99)00263-x. PMID 10389720
- [Background] Lemack GE, Zimmern PE. Predictability of urodynamic findings based on the Urogenital Distress Inventory-6 questionnaire. Urology. 1999 Sep;54(3):461-6. doi: 10.1016/s0090-4295(99)00246-0. PMID 10475355
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Eisenstein SM, Engelbrecht DJ, el Masry WS. Low back pain and urinary incontinence. A hypothetical relationship. Spine (Phila Pa 1976). 1994 May 15;19(10):1148-52. doi: 10.1097/00007632-199405001-00010. PMID 8059271
- [Background] Shumaker SA, Wyman JF, Uebersax JS, McClish D, Fantl JA. Health-related quality of life measures for women with urinary incontinence: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res. 1994 Oct;3(5):291-306. doi: 10.1007/BF00451721. PMID 7841963
- [Background] Minaire P, Jacquetin B. [The prevalence of female urinary incontinence in general practice]. J Gynecol Obstet Biol Reprod (Paris). 1992;21(7):731-8. French. PMID 1469226
- [Background] Norton PA, MacDonald LD, Sedgwick PM, Stanton SL. Distress and delay associated with urinary incontinence, frequency, and urgency in women. BMJ. 1988 Nov 5;297(6657):1187-9. doi: 10.1136/bmj.297.6657.1187. No abstract available. PMID 3144344
- [Background] Thom D. Variation in estimates of urinary incontinence prevalence in the community: effects of differences in definition, population characteristics, and study type. J Am Geriatr Soc. 1998 Apr;46(4):473-80. doi: 10.1111/j.1532-5415.1998.tb02469.x. PMID 9560071
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Tsao H, Hodges PW. Immediate changes in feedforward postural adjustments following voluntary motor training. Exp Brain Res. 2007 Aug;181(4):537-46. doi: 10.1007/s00221-007-0950-z. Epub 2007 May 3. PMID 17476489